CLINICAL TRIAL: NCT06252246
Title: The Effect of Phacoemulsification on Intraocular Pressure in Primary Angle Closure Glaucoma (PACG) Patients At Phanat Nikhom Hospital, Chonburi Province
Status: Completed | Type: Observational
Sponsor: Phanatnikhom Hospital (Other Government)
Responsible Party: Principal Investigator, Thetthar Kanthar, Head of Ophthalmology, Ophthalmological department, Phanatnikhom Hospital
Other Study IDs: 5100500081212
Record Dates: First submitted 2024-01-20; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Primary Angle Closure Glaucoma
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Phacoemulsification machine — type of phacoemulsification machine is different

SUMMARY:
BACKGROUND: Primary angle closure glaucoma (PACG) is one of a leading cause of blindness worldwide including Thailand. This problem impact to the overall health of people and health care system. Treatment guidelines of each stage is differenced. Therefore, factors that affect to treatment should be explored to plan for taking care patients in the future.

OBJECTIVES: The study aimed to examine the effects of cataract surgery by phaco- emulsification on intraocular pressure and to determine the factors associated with intraocular pressure among primary angle closure glaucoma patients.

DETAILED DESCRIPTION:
BACKGROUND: Primary angle closure glaucoma (PACG) is one of a leading cause of blindness worldwide including Thailand. This problem impact to the overall health of people and health care system. Treatment guidelines of each stage is differenced. Therefore, factors that affect to treatment should be explored to plan for taking care patients in the future.

OBJECTIVES: The study aimed to examine the effects of cataract surgery by phaco- emulsification on intraocular pressure and to determine the factors associated with intraocular pressure among primary angle closure glaucoma patients.

METHODS: A retrospective descriptive study was conducted in 121 patients with primary angle closure glaucoma who underwent phacoemulsification between October 1st 2017 and September 30th 2022. The preoperative and postoperative record form were used as the research instrument. Visual acuity, intraocular pressure, the number of glaucoma medications and ocular biometric parameters were collected. The descriptive statistics, Paired sample t-test, Repeated measures ANOVA and Multiple linear regression were used to analyze the outcomes. A p-value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age more 18 years old and not complication of cataract surgey

Exclusion Criteria:

* other eye diseases affect to visual defect
* previous ocular surgery
* complication of cataract surgery
* data record incomplete

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary angle closure glaucoma (PACG) is one of a leading cause of blindness worldwide including Thailand. This problem impact to the overall health of people and health care system. Treatment guidelines of each stage is differenced. Therefore, factors that affect to treatment should be explored to plan for taking care patients in the future
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
intraocular pressure | six months
  effects of cataract surgery by phacoemulsification on intraocular pressure and to determine the factors associated with intraocular pressure among primary angle closure glaucoma patients. Units of measure assessment intraocular pressure by non contact tonometry(intraocular pressure in millimeters of Mercury) at one week, one month, three months and six months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Phanatnikhom hospital, Chon Buri, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Undecided